CLINICAL TRIAL: NCT00825045
Title: Dopamine D2 and D3 Receptor Occupancy and Clinical Response in Older Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Ariel Graff, MD, PhD, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 270/2008
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: dopamine; D2; D3; caudate; putamen; globus pallidus; antipsychotic; risperidone; geriatric; Brief Psychiatric Rating Scale; PET; radiotracer; [11C]-(+)-PHNO; [11C]-raclopride
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with risperidone (Experimental): Gradual titration of risperidone according to clinical response
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: risperidone — Following the baseline clinical and cognitive assessments, risperidone will be initiated at 0.5-1.0 mg/day and subsequently increased by 0.25 - 1.0 mg on a weekly basis with the target of clinical stabilization (i.e. 20 or more % reduction in the total BPRS score) until a maximum dose of 4.0 mg/day is reached. To achieve this, a weekly assessment with BPRS will be performed. Physicians-of-record will be closely liaised with investigators. Dosage modification will be performed following this dosing schedule, however, this can be changed by treating physicians to meet clinical necessity. For example, in case psychotic symptoms are not controlled by this dosing schedule, facilitated dose increment will be allowed.

SUMMARY:
This study will provide information regarding dopamine D2/D3 occupancy related with clinical/adverse effects in older people with schizophrenia and schizoaffective disorder. The results of this study will also show an appropriate dose range in order to evade undesirable adverse effects while deriving therapeutic effects, which will directly serve to guide physicians in clinical practice. Furthermore, the findings of this study will elucidate mechanisms underlying older people's increased sensitivity to antipsychotic drugs. In addition, the contribution of D2 and D3 in mediating antipsychotic response will be contrasted, using 2 radiotracers, which has never been tested in an older population.

The hypotheses are as follows: First, clinical response (i.e., a ≥ 20% decrease in the Brief Psychiatric Rating Scale total score) will be achieved in older patients with occupancy that is lower than the threshold of 60% in historical young controls. Second, prolactin elevation and EPS will be detected in older patients with occupancies that are lower than the thresholds of 72 and 78% reported in historical young controls. Third, dopamine D2 receptor occupancy will be inversely correlated with subjective well-beings. Fourth, the binding potential and receptor occupancy will be at least 20% lower with [11C]-(+)-PHNO than with [11C]-raclopride in the caudate/putamen. Fifth, the binding of [11C]-(+)-PHNO in the globus pallidus will be higher than that of [11C]-raclopride.

DETAILED DESCRIPTION:
Positron Emission Tomography (PET) studies have demonstrated that a therapeutic window of dopamine D2/3 receptor occupancy (60-80%) is associated with clinical response in younger patients with schizophrenia. This observation has been used to predict the therapeutic dose range and contributed to current recommended antipsychotic doses. To date, there is no published report to examine D2/3 receptor occupancy associated with clinical response in older individuals with primary psychotic disorders. This has has impeded the implementation of treatment guidelines.

The investigators therefore propose a prospective study to assess dopamine D2 and D3 receptor occupancy following acute antipsychotic treatment in patients aged 50 and older with schizophrenia who do not currently receive antipsychotic treatment, using both [11C]-(+)-PHNO and [11C]-raclopride PET scans. Dopamine D2/3 receptor occupancy of risperidone that are associated with clinical effects will be measured, using PET, in older patients with schizophrenia. The investigators will also try to contrast the contribution of D2 and D3 in mediating antipsychotic response, using 2 radiotracers.

Our primary goal is to relate changes in clinical outcome, including subjective and objective clinical ratings, to dopamine D2 and D3 receptor occupancy in older patients with schizophrenia, and compare these results with the data for younger patients in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Age of 50 and older at time of scanning
* Inpatients or outpatients
* DSM-IV/SCID diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorder
* Having NOT been treated with oral antipsychotic treatment for at least 2 weeks or long-acting antipsychotics for at least 6 months (Please note that patients will not be withdrawn from antipsychotic medications for the purpose of meeting inclusion criteria for this study).

Exclusion Criteria:

* Known history of intolerance or inefficacy to risperidone
* Participation in this study would result in exceeding the annual radiation dose limits (20 mSv) for human subjects participating in research studies.
* Substance abuse or dependence (within past six months)
* Positive urine drug screen
* Positive serum pregnancy test at screening or positive urine pregnancy test before PET scan
* Metal implants or a pace-maker that would preclude the MRI scan
* History of head trauma resulting in loss of consciousness >30 minutes that required medical attention
* Unstable physical illness or significant neurological disorder including a seizure disorder
* Inappropriate size of head, neck, and body to be able to fit the PET and MRI scans

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2008-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The occupancy of risperidone at the D2 and D3 receptor, using [11C]-raclopride and [11C]-(+)-PHNO, respectively. | Within 3 months of enrollment

SECONDARY OUTCOMES:
Plasma levels of risperidone and 9-hydroxyrisperidone | Within 3 months of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Graff-Guerrero, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research